CLINICAL TRIAL: NCT05061641
Title: Study on the Prediction and Prevention of Twin Premature Birth
Brief Title: Prediction and Prevention of Twin Premature Birth 2021
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Caixia Liu (Other)
Responsible Party: Sponsor-Investigator, Caixia Liu, Shengjing hospital, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPB 2021
Record Dates: First submitted 2021-06-26; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Who Masked: Participant, Care Provider
Masking Description: The participants and the treating physicians were not informed of the grouping
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- progesterone 200mg (Active Comparator): Each group was given prophylactic vaginal progesterone up to 34 weeks of gestation，Vaginal progesterone 200mg
  Interventions: Drug: Progesterone
- progesterone 400mg (Experimental): Each group was given prophylactic vaginal progesterone up to 34 weeks of gestation，Vaginal progesterone 400mg
  Interventions: Drug: Progesterone
- progesterone 600mg (Experimental): Each group was given prophylactic vaginal progesterone up to 34 weeks of gestation，Vaginal progesterone 600mg
  Interventions: Drug: Progesterone

INTERVENTIONS:
Drug: Progesterone — The delivery outcomes of the three groups were compared, including the rate of premature delivery (<37 weeks of gestation), the rate of early premature delivery (<32 weeks of gestation), and the need for anti-tocolysis treatment. Rates of premature rupture of membranes (<37 weeks), neonatal perinatal mortality and morbidity.
  Other Names: surgical treatment

SUMMARY:
Research Objectives:

1. Establish a prediction and scoring system for twin premature birth.
2. To investigate the curative effect of 200mg,400mg and 600mg of vaginal progesterone in the prevention of twin premature birth.
3. To investigate the effect of stress cervical ligation in preventing premature delivery of twins.
4. The optimal dose of atosiban for the treatment of twin premature birth.
5. The influence of delivery mode on twin premature infants under 32 weeks.

DETAILED DESCRIPTION:
Research Objectives:

1. Establish a prediction and scoring system for twin premature birth.
2. To investigate the curative effect of 200mg,400mg and 600mg of vaginal progesterone in the prevention of twin premature birth.
3. To investigate the effect of stress cervical ligation in preventing premature delivery of twins.
4. The optimal dose of atosiban for the treatment of twin premature birth.
5. The influence of delivery mode on twin premature infants under 32 weeks. It has now entered the second phase: clinical data collection

ELIGIBILITY:
Inclusion Criteria:

twins with cervical length ≤ 25 mm by vaginal ultrasound at 14-32 weeks no contractions, abdominal pain and vaginal bleeding No complicated twin complications occurred during pregnancy

Exclusion Criteria:

Patients undergoing selective cervical ligation before 14 weeks of gestation history of liver problems or cholestasis during pregnancy Abnormal liver enzymes Abnormal renal function Local allergy to trace natural progesterone Recurrent vaginal bleeding Recurrent vaginal infection Ultrasound diagnosis of fetal abnormality Intrauterine treatment for fetal abnormalities

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Neonatal prognosis | one week
  Preterm birth rate (<37 weeks of gestation), early preterm birth rate (<32 weeks of gestation), need to receive anti-tocolytic treatment; Rates of premature rupture of membranes (<37 weeks), neonatal perinatal mortality and morbidity.

SECONDARY OUTCOMES:
Gestational age and prolongation of gestational age at delivery | one year
  Gestational age at which symptoms of preterm birth occur and gestational age at delivery after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wei jun, Dr, Study Chair — 1050880483@qq.com
Locations (1):
- caixia Liu, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No